CLINICAL TRIAL: NCT05237869
Title: Blood Flow Restricted Training to Enhance Lateral Epicondylitis Rehabilitation.
Brief Title: Blood Flow Restriction & Tennis Elbow Rehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Nuelle (Other)
Responsible Party: Sponsor-Investigator, Julie Nuelle, Assistant Professor of Orthopaedic Surgery, Hand Surgeon, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2070985
Record Dates: First submitted 2021-12-27; First posted 2022-02-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: For patients enrolled in the control group, the participants will undergo calibration of the Delfi Personalized Tourniquet System to measure limb occlusion pressure and will wear the cuff during completion of the exercises with minimal inflation (approximately 5%), to hold the cuff in place during treatment. This will act as a sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Physical Therapy (Sham Comparator): For patients enrolled in the control group, the participants will undergo calibration of the Delfi Personalized Tourniquet System to measure limb occlusion pressure and will wear the cuff during completion of the exercises with minimal inflation (approximately 5%), to hold the cuff in place during treatment. This will act as a sham.
  Interventions: Other: Standard Physical Therapy
- Blood Flow Restricted Physical Therapy (Active Comparator): Physical therapy assisted by blood flow restriction per standard physical therapy protocol.
  Interventions: Device: Blood Flow Restriction Device

INTERVENTIONS:
Device: Blood Flow Restriction Device — Occlusion training involves the application of a cuff to the upper arm that is designed to restrict only the low-pressure blood flow in veins. It does not prevent blood flowing from the heart to the arm.
  Arms: Blood Flow Restricted Physical Therapy
Other: Standard Physical Therapy — Standard physical therapy protocol for lateral epicondylitis rehab without blood flow restriction.
  Arms: Physical Therapy

SUMMARY:
Lateral epicondylitis (LE), often referred to as "tennis elbow" is a common and debilitating overuse injury affecting 1-3% of adults annually. LE is most often defined as a syndrome of pain near the area of the lateral epicondyle of the elbow commonly effecting the origin of the extensor carpi radialis brevis with associated weakness; it most commonly effects the dominant arm. The best treatment for LE is unknown and research to support current treatment methods are insufficient. A common limitation in functional recovery experienced by this population is pain at the lateral aspect of the elbow. As such, innovative therapeutic interventions directed at quickly reducing pain may address this unmet need and allow for improved outcomes, as well as earlier return to function.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65 years of age
2. Diagnosis of lateral epicondylitis confirmed by the treating orthopaedic surgeon and ultrasound
3. Must be able to read and write in English
4. Able to provide own written consent

Exclusion Criteria:

1. Patients over 65 years of age
2. Contralateral upper extremity involvement resulting in less than normal range of motion, muscle strength or daily pain greater than 1/10
3. History of prior injection for treatment of lateral epicondylitis
4. Pregnancy
5. Recent history of deep venous thrombosis (within the past 12 months)
6. Active treatment with anticoagulants
7. History of upper quadrant lymph node dissection
8. History of endothelial dysfunction
9. Patient history of easy bruising
10. Active infection in the injured arm
11. Cancer
12. Uncontrolled peripheral vascular disease
13. Uncontrolled diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Define the effect of BFR training on pain with activity in patients with LE. | 3 weeks to 6 months
  Measured on a 0-10 scale by VAS (Visual Analog Scale) patient reported outcome form. The VAS is scored 0-10, and a higher score indicates worse pain/worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Nuelle, MD, Principal Investigator — University of Missouri Department of Orthopaedic Surgery
Locations (1):
- Vicki Jones, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No